CLINICAL TRIAL: NCT01205321
Title: Open-label, Multi Center PET/CT (Positron Emission Tomography/Computed Tomography) Study for Investigation of Safety, Tolerability, Biodistribution and Diagnostic Performance of the 68Ga Labeled PET Tracer BAY86-7548 Following a Single Intravenous Administration of 140 MBq (Corresponding to ≤ 28 µg Mass Dose) in Patients With Prostate Cancer as Well as Radiation Dosimetry, Plasma Pharmacokinetics, Biodistribution, Safety and Tolerability of the Tracer in PET/CT in Healthy Volunteers
Brief Title: PET/CT Imaging for Radiation Dosimetry, Plasma Pharmacokinetics, Biodistribution, Safety and Tolerability and Diagnostic Performance of BAY86-7548 in Patients With Prostate Cancer and Healthy Volunteers
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: Life Molecular Imaging SA (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Diagnostic
Other Study IDs: 14269; 2008-008315-25 (EudraCT Number)
Record Dates: First submitted 2010-09-17; First posted 2010-09-20 (Estimated); Last update posted 2013-01-21 (Estimated); Status verified 2013-01

CONDITIONS: Diagnostic Imaging
Keywords: Neoplasm; PET/CT diagnosis; PET tracer
MeSH Terms: conditions — Neoplasms | interventions — Bombesin; Product Labeling; BAY 86-7548

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (2):
- Arm 1 (Experimental)
  Interventions: Drug: Bombesin (68Ga) labeled (BAY86-7548)
- Arm 2 (Experimental)
  Interventions: Drug: Bombesin (68Ga) labeled (BAY86-7548)

INTERVENTIONS:
Drug: Bombesin (68Ga) labeled (BAY86-7548) — Cancer patients, single intravenous bolus injection of 140 MBq BAY86-7548 on day one of the treatment period, PET/CT
  Arms: Arm 1
Drug: Bombesin (68Ga) labeled (BAY86-7548) — Healthy volunteers, single intravenous bolus injection of 140 MBq BAY86-7548 on day one of the treatment period, whole body PET/CT for determination of effective dose, kinetics of BAY86-7548 in blood
  Arms: Arm 2

SUMMARY:
Visual assessment of diagnostic PET/CT (positron emission tomography/computed tomography) images obtained after a single intravenous injection of BAY86-7548 in patients with cancer.

ELIGIBILITY:
Inclusion Criteria:

* Healthy volunteers:

  * males, >/=50 and </= 65 years of age
* Cancer patients:

  * males >/= 45 years of age
  * Patients had an MRI of the prostate and/or a positive choline or acetate PET/CT for diagnosis (Note: MRI, choline and acetate PET/CT are optional for primary prostate cancer patients) of recurrence prostate cancer and the primary cancer disease is/ will be histologically confirmed.
  * The prostate cancer is histologically confirmed and results of histology are available.
  * Patients with primary prostate cancer: >/= 20 percent of biopsy material should be affected by cancer in the histopathological evaluation.
  * Patients with primary prostate cancer: Patient is scheduled to undergo prostatectomy.

Exclusion Criteria:

* Concurrent severe and/or uncontrolled and/or unstable other medical disease (e.g. poorly controlled diabetes, congestive heart failure, myocardial infarction within 12 months prior to planned injection of BAY86-7548, unstable and uncontrolled hypertension, chronic renal or hepatic disease, severe pulmonary disease) which could compromise participation in the study
* Known sensitivity to the study drug or components of the preparation.

Min Age: 45 Years | Sex: Male | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 19 (Actual)
Dates: Start 2010-11; Primary Completion 2011-11 (Actual); Study Completion 2011-12 (Actual)

PRIMARY OUTCOMES:
Visual assessment of lesions | Day of study drug administration

SECONDARY OUTCOMES:
Quantitative analysis of BAY86-7548 uptake into lesions (Standardized Uptake Values = SUVs) | Day of study drug administration
ECG (significant abnormalities) | At least 3 times until one day after treatment
Blood pressure | At least 3 times until one day after treatment
Serum protein | At least 3 times until one day after treatment
Serum creatinine | At least 3 times until one day after treatment
Serum GOT (Glutamat-Oxalacetat-Transaminase) | At least 3 times until one day after treatment
Adverse events collection | Continuously for at least 5 days after treatment

CONTACTS AND LOCATIONS:
Overall Officials: Bayer Study Director, Study Director — Bayer
Locations (3):
- Turku, Finland
- Ulm, Baden-Wurttemberg, Germany
- Zurich, Canton of Zurich, Switzerland